CLINICAL TRIAL: NCT06006000
Title: Evaluating the Unmet Needs of Older Adults to Promote Functional Recovery After a Critical Illness
Acronym: LANTERN
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2000034943; 1R01AG079916-01A1 (NIH)
Record Dates: First submitted 2023-08-15; First posted 2023-08-23 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Critical Illness; Illness, Critical
Keywords: Geriatrics; Older Adults
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adults returning home post-ICU: Community-dwelling older adults who return home (either directly or after a stay in short-term rehab (STR)) after an ICU hospitalization.

SUMMARY:
This is a prospective longitudinal study that will evaluate the unmet needs of older adults (65 and older) who return home (either directly or after short-term rehab) after an ICU hospitalization, evaluate the association of these unmet needs with clinically relevant outcomes, and assess barriers and facilitators to addressing these unmet needs. The proposed research will inform the development and evaluation of a subsequent intervention to improve functional outcomes among older ICU survivors, in alignment with the NIH's mission to reduce disability.

DETAILED DESCRIPTION:
To identify unmet needs in multiple domains after return home from an ICU hospitalization, evaluate whether these unmet needs are associated with disability burden in the subsequent 6 months, and ascertain whether these associations are moderated by initial discharge destination (home or STR).

ELIGIBILITY:
Inclusion Criteria:

PARTICIPANTS

* Age ≥ 65 years
* Survived an ICU admission of ≥2 days

CAREGIVERS

* Age ≥ 18 years
* Identified as caregiver of LANTERN participant who is an informal (unpaid) caregiver.

Exclusion Criteria:

PARTICIPANTS

* Advance directive of comfort measures only (CMO) or a transition to hospice
* Planned discharge to a location other than home or Short-Term Rehab
* Tracheostomy with ventilator dependence
* Severe acute or prior neurologic injury (such as anoxic brain injury or acute, massive stroke)
* Advanced dementia
* ICU admission for monitoring only (e.g., antibiotic desensitization)
* Primary language other than English.
* Homelessness
* Active drug or alcohol use disorder.

CAREGIVERS

* Primary language other than English
* Is a paid caregiver
* Unwilling to complete a qualitative interview

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Community-dwelling older adults who return home (either directly or after a stay in short-term rehab (STR)) after an ICU hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Disability Count | monthly up to 6 months
  Number of instances of disability during activities of daily living (ADLs), instrumental activities of daily living (IADLs), and mobility activity. Disability is defined as an inability to complete the task or the need for personal assistance to complete the task. The higher the count, the more disability.
Number of hospital readmissions | monthly up to 6 months
  Number of hospital readmissions monthly up to 6 months.
Number of deaths | monthly up to 6 months
  Number of deaths each month up to 6 months.
Barriers and Facilitators to addressing unmet needs | month 6
  Barriers and facilitators to addressing unmet needs will be assessed using qualitative interviews. A subgroup of participants will receive qualitative interviews conducted with members of the study team. Content analysis will then be used to identify barriers and facilitators to addressing unmet needs that will be informative when planning a future intervention.

SECONDARY OUTCOMES:
Functional non-recovery | monthly up to 6 months
  Not returning to the pre-ICU functional baseline within the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Ferrante, MD, MHS, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data from this study will be available to investigators who sign a Data Use Agreement (DUA) executed between Yale University and the investigator's institution. The DUA requires the investigators to attest to (1) their commitment to using the data only for approved research purposes and not to identify any individual human participant; (2) their commitment to securing the data using appropriate computer technology; and (3) their commitment to destroying or returning the data after analyses are completed.
  Data will not be available until all analyses are complete.